CLINICAL TRIAL: NCT00820417
Title: Phase 1 Pharmacokinetic (PK) and Pharmacodynamic (PD) Study of the Combination of Cetuximab (C-225), a Chimeric Monoclonal Antibody Against the Epidermal Growth Factor Receptor (EGFR), and Gefitinib (ZD1839), a Selective EGFR Tyrosine Kinase Inhibitor, in Patients With Advanced Cancer
Brief Title: Pharmocokinetic/Pharmacodynamic (PK/PD) Study of the Combination Cetuximab/Gefitinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Harrison Clinical Research (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry); AstraZeneca (Industry)
Responsible Party: Josep Tabernero, MD, Head, Gastrointestinal Cancer Unit, Medical Oncology Department, Vall d'Hebron University Hospital
Allocation: Non-Randomized | Masking: None
Other Study IDs: C-225/ZD1839
Record Dates: First submitted 2009-01-09; First posted 2009-01-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Colorectal Cancer; Head and Neck Cancer; Non Small Cell Lung Cancer (NSCLC)
Keywords: cetuximab; monoclonal; antibody; epidermal; growth; factor; receptor; EGFR; Gefitinib; tyrosine; kinase; inhibitor; advanced; cancer
MeSH Terms: conditions — Colorectal Neoplasms; Head and Neck Neoplasms; Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- a (Experimental): Dose-escalation
  Interventions: Drug: Cetuximab/Gefitinib combination and/or monotherapy
- B (Experimental): Maximum tolerated dose (MTD)
  Interventions: Drug: Cetuximab/Gefitinib combination and/or monotherapy

INTERVENTIONS:
Drug: Cetuximab/Gefitinib combination and/or monotherapy

SUMMARY:
This is an open-label, phase 1, non-randomised, non-controlled trial, carried out in two centres on patients with advanced cancer expressing EGFR. Primary objective is the determination of the maximum tolerated dose (MTD) and recommended dose (RD) of the combination of intravenous Cetuximab and oral Gefitinib.

DETAILED DESCRIPTION:
Between 36 and 66 patients will be enrolled depending on the number of dose levels which can be completed. Patients will have histologically confirmed EFGR-expressing solid malignant tumours (colorectal cancer, head and neck cancer and NSCLC), which did not respond to standard therapy or for which no suitable therapy exists.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent prior to inclusion
* Confirmed histological diagnosis of non-resectable, solid, malignant, EGFR expressing tumours of the following types: colorectal cancer, head and neck cancer and non-small cell lung cancer (NSCLC). Advanced clinical stage III/IV which did not respond to standard therapy or for which no suitable therapy exists
* Patients with at least one evaluable lesion (evaluable disease) by the RECIST criteria
* Availability of tumour tissue, whether from primary tumour or metastasis to determine EGFR expression
* Viability of establishing outpatient treatment
* Effective contraception for patients of both sexes if there is a risk of conception
* Karnofsky performance status greater than 70 %
* Life expectancy > 12 weeks
* Adequate renal function (creatinine < 1.5 x UNL), liver function (bilirubin < 1.5 x UNL, ALT/AST < 2.5 x UNL o <5 x UNL if hepatic metastasis) and adequate bone marrow (leucocytes > 3000/µl, absolute neutrophil count > 1500/µl, platelets > 100,000/µl, haemoglobin > 9 g/dl)
* Patients must not have undergone chemotherapy, radiotherapy or major surgery during the 3 weeks before the beginning of the study, and they must have recovered from the relevant secondary effects of previous treatments
* Patients agree to have a new biopsy after two weeks.

Exclusion Criteria:

* Patients with any symptom of bowel obstruction and/or inflammatory bowel disease
* Previous therapy with anti-EGFR drugs
* Patients with known cerebral metastasis
* Patients with known active and uncontrolled infections
* Severe uncontrolled organic dysfunctions or metabolic disorders
* Patients unable to give informed consent
* Patients who do not wish to or who cannot undergo the specific study treatments and the study procedures
* Pregnancy or breastfeeding
* Patient participation in another clinical trial during the previous 30 days
* Patients with known drug and/or alcohol abuse
* Known hypersensitivity to chimeric MoAbs or pretreatment with MoAbs
* Any other malignant tumour in the last two years or previously diagnosed malignant tumour if there is no guarantee that it is under complete control, except for suitably treated in situ cervical carcinoma or basocellular carcinoma
* Known severe hypersensitivity to ZD1839 or any of the excipients of this product
* Any evidence of clinically active interstitial lung disease (patients with chronic, stable, radiographic changes who are asymptomatic need not to be excluded)
* Any unresolved chronic toxicity greater than common toxicity criteria (CTC) grade 2 from previous anticancer therapy
* Concomitant use of phenytoin, carbamazepine, rifampicin, barbiturates, or St John's Wort

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2004-06; Primary Completion 2007-09 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The primary objective of the study is to determine the maximum tolerated dose (MTD) and the recommended dose (RD) of the combination intravenous Cetuximab/oral Gefitinib.

SECONDARY OUTCOMES:
To determine the pharmacokinetic (PK) parameters of the combination Cetuximab/Gefitinib
To determine the pharmacogenomic profile of study patients and to correlate the different profiles with efficacy
To determine the possible correlation between activity and the polymorphisms of the EGFR measured in the blood and in the primary tumour
To assess the possible immune response related to cetuximab
To estimate signs of clinical activity (response rate according to the RECIST criteria)

CONTACTS AND LOCATIONS:
Locations (2):
- UZ Gasthuisberg, Leuven, Belgium
- Hospital Universitari Vall d'Hebron, Barcelona, Spain